CLINICAL TRIAL: NCT00578019
Title: Prospective Comparison Between Less Invasive Stabilization System (LISS) Plating and Intramedullary Nailing for the Treatment of Supracondylar Femur Fractures
Brief Title: Comparison Between LISS Plating and Intramedullary (IM) Nailing for Supracondylar Femur Fractures
Acronym: LISS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: James P. Stannard, MD, Professor of Surgery, Assoc. Director of Orthopaedic Surgery, The University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F990825010; AO Foundation FORK 99S83
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Supracondylar Femur Fracture
Keywords: Comparative; Supracondylar Femur Fracture; Intramedullary nailing; Less Invasive Stabilization System (LISS) Plating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1, A (Active Comparator)
  Interventions: Procedure: IM Nailing
- 2, B (Experimental): Group B patients will have their fracture stabilized with the LISS plates (Synthes [USA], Paoli, PA, USA).
  Interventions: Procedure: LISS

INTERVENTIONS:
Procedure: IM Nailing — Patients randomized to Arm 1, A will be treated with a retrograde intramedullary nailing of the femur fracture utilizing the Smith & Nephew supracondylar nail.
  Other Names: Smith & Nephew Supracondylar Nail
  Arms: 1, A
Procedure: LISS — Group B patients will have their fracture stabilized with the LISS plates (Synthes [USA], Paoli, PA, USA).
  Other Names: Synthes LISS
  Arms: 2, B

SUMMARY:
The purpose of this study is to compare patient outcomes for the Less Invasive Stabilization System (LISS) (Synthes {USA}, Paoli, PA, USA), a minimally invasive plating system used in the treatment of supracondylar femur fractures, with patient outcomes for the Supracondylar Nail (Smith & Nephew Inc, Memphis, TN, USA), a retrograde intramedullary nail.

DETAILED DESCRIPTION:
All patients who meet the inclusion and exclusion criteria will be randomized into one of two treatment groups. Group A patients will be treated with retrograde intramedullary nailing of the fracture with supplemental screw fixation of the articular portion of the fracture if needed. The Richards supracondylar nail (Smith & Nephew Richards, Memphis, TN, USA) will be utilized. Group B patients will have their fracture stabilized with the LISS plates (Synthes [USA], Paoli, PA, USA). Supplemental screw fixation of the articular portion of the fracture will occur, if needed. Postoperative care will not be any different than the postoperative care of any other patient undergoing internal fixation of a complex fracture around the knee and based on the patient's overall condition.

Surgical Protocol: After the anesthesia staff has administered general anesthesia, the patient will be positioned on the operating room table as described by the intraoperative technique guide or according to the patient's injury and the surgeon's preference. The patient will be prepped and draped in the usual and customary manner for orthopaedic procedures of the lower extremities. The image intensifier will be available for intraoperative fluoroscopy. The manufacturer's surgical technique guide will be used intraoperatively for implantation of the LISS device and the supracondylar nail. The surgical wound will be closed according to the surgeon's preference. A drainage device may be used if indicated. Routine dressings will be applied. In all instances, immediate postoperative radiographs will be taken to document adequate reduction and fixation. Neurovascular evaluation of the extremity will be performed and documented when the patient emerges from the anesthetic. The patient will be discharged from the recovery room to the postoperative unit when they have met discharge criteria. Routine postoperative orders will be followed until discharge from the hospital.

Patients will be followed in the orthopaedic clinic at predetermined intervals following surgery. The clinic visits will include anterior-posterior and lateral radiographs of the affected extremity and a clinical examination. The patient will also complete the SF-36 (Appendix 1) and a pain scale (Appendix 2). This data will be used to compare the outcomes obtained with the two devices. Clinical follow-up will occur at 2, 4, 8, 12, 18, 26, and 52 weeks following surgery. Radiographs will be obtained at 4, 8, 12, 18, 26, and 52 weeks postoperatively. Patients will complete pain scales at 4, 8, 12, 18, 26, and 52 weeks after surgery. Clinical outcomes will be evaluated at weeks 12, 26, and 52.

ELIGIBILITY:
Inclusion Criteria:

* Type A or C supracondylar femur fracture
* Adult patients (19 years or older)

Exclusion Criteria:

* Patients unable or unwilling to comply with follow-up gait, radiographic, and clinical evaluations necessary to complete the study
* Patients are not able or willing to give informed consent and/or have no responsible family member willing to give consent
* Patients with a disease entity or condition that totally precludes the possibility of bony fusion or patients undergoing drug therapy that prevents bony healing
* Mentally retarded persons
* Mentally disabled individuals
* Prisoners
* Pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 1999-12; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is complete healing of the femur fracture | Clinical outcomes will be evaluated at weeks 12, 26, and 52

SECONDARY OUTCOMES:
Secondary outcome is to compare the time and quality of healing of the femur fracture | Will be evaluated at weeks 12, 26 and 52

CONTACTS AND LOCATIONS:
Overall Officials: James P Stannard, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Orthopaedic Trauma, Birmingham, Alabama, United States

REFERENCES:
- [Background] Kayali C, Agus H, Turgut A. Successful results of minimally invasive surgery for comminuted supracondylar femoral fractures with LISS: comparative study of multiply injured and isolated femoral fractures. J Orthop Sci. 2007 Sep;12(5):458-65. doi: 10.1007/s00776-007-1156-8. Epub 2007 Sep 28. PMID 17909931
- [Background] Boldin C, Fankhauser F, Hofer HP, Szyszkowitz R. Three-year results of proximal tibia fractures treated with the LISS. Clin Orthop Relat Res. 2006 Apr;445:222-9. doi: 10.1097/01.blo.0000203467.58431.a0. PMID 16456310
- [Background] Stannard JP, Wilson TC, Volgas DA, Alonso JE. The less invasive stabilization system in the treatment of complex fractures of the tibial plateau: short-term results. J Orthop Trauma. 2004 Sep;18(8):552-8. doi: 10.1097/00005131-200409000-00012. PMID 15475852